CLINICAL TRIAL: NCT01164228
Title: A Randomized Phase II Trial of Sunitinib/Gemcitabine or Sunitinib in Advanced Renal Cell Carcinoma With Sarcomatoid Features
Brief Title: Sunitinib Malate With or Without Gemcitabine Hydrochloride in Treating Patients With Advanced Kidney Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E1808; NCT01164228 (Registry Identifier: ClinicalTrials.gov); NCI-2011-02055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA021115 (NIH)
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma; papillary renal cell carcinoma; clear cell sarcoma of the kidney
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gemcitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Sunitinib + Gemcitabine) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 22, and 29 and oral sunitinib malate once daily on days 1-14 and 22-35. Each cycle was 42 days (6 weeks) and was to be repeated for a total of one year.
  Interventions: Drug: Gemcitabine; Drug: Sunitinib
- Arm B (Sunitinib) (Experimental): Patients receive oral sunitinib malate once daily on days 1-14 and 22-35. Each cycle was 42 days (6 weeks) and was to be repeated for a total of one year.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: 2'-Deoxy-2'; 2'-difluorocytidine monohydrochloride; Gemzar
  Arms: Arm A (Sunitinib + Gemcitabine)
Drug: Sunitinib — Given PO
  Other Names: SU011248 L-Malate salt; SU010398; PHA-290940AD; Sutent; SU011248

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth or tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving sunitinib malate and gemcitabine hydrochloride together is more effective than sunitinib malate alone in treating patients with kidney cancer.

PURPOSE: This randomized phase II clinical trial is studying giving sunitinib malate together with or without gemcitabine hydrochloride to see how well they work in treating patients with advanced kidney cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the response rate to sunitinib malate with vs without gemcitabine hydrochloride in patients with advanced renal cell carcinoma with sarcomatoid features.

Secondary

* To evaluate progression-free survival of these patients.
* To evaluate overall survival of these patients.
* To describe the toxic effects of both sunitinib malate alone and in combination with gemcitabine hydrochloride in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to risk (good risk [clear cell and < 20% sarcomatoid and performance status (PS) 0] vs intermediate risk [20-50% sarcomatoid and PS 0] vs poor risk [non-clear cell or > 50% sarcomatoid or PS 1 or non-clear cell]). Patients are randomized to 1 of 2 treatment arms.

* Arm A: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, 22, and 29 and oral sunitinib malate once daily on days 1-14 and 22-35.
* Arm B: Patients receive oral sunitinib malate once daily on days 1-14 and 22-35.

In both arms, courses repeat every 42 days for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 1 year.

ACTUAL ACCRUAL: A total of 87 patients (47 in arm A and 40 in arm B) were accrued to this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed* renal cell carcinoma of any subtype containing any sarcomatoid features NOTE: *Patients must have a paraffin-embedded tumor specimen from the kidney or metastatic site available for central review and confirmation of tumor histology
* Measurable advanced disease that is not resectable by surgery
* Patients with resected or radiated brain metastases or those treated with stereotactic radiation therapy are eligible, provided they have been off steroids for at least 2 weeks
* More than 2 weeks since prior radiotherapy and recovered

  * Previously irradiated lesions must not be the sole site of disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL (transfusions allowed)
* Serum creatinine clearance ≥ 30 mL/min
* serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 times upper limit of normal (ULN; ≤ 5 times ULN in the presence of liver metastases)
* Total bilirubin ≤ 1.5 times ULN
* Baseline corrected QT interval < 500 msec on EKG
* Able to swallow pills
* Negative pregnancy test
* Fertile patients must use effective contraception before and during study treatment
* More than 2 weeks since prior and no concurrent ketoconazole, dexamethasone, dysrhythmic drugs (terfenadine, quinidine, procainamide, sotalol, probucol, bepridil, indapamide, or flecainide), haloperidol, risperidone, rifampin, grapefruit, or grapefruit juice
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been disease free for the time period considered appropriate to not interfere with the outcome of this study

Exclusion Criteria:

* Collecting duct or medullary carcinoma
* Prior systemic therapy for metastatic disease. One prior therapeutic regimen with a non-tyrosine kinase inhibitor, such as an mtor inhibitor is allowed. Patients who were randomized to placebo on an adjuvant study are eligible
* History of stroke within the past 6 months.
* Pregnant or nursing
* Clinically significant cardiovascular disease, defined as one of the following:

  * Uncontrolled hypertension (blood pressure > 150/100 mm Hg at the time of enrollment); patients with hypertension and BP ≤ 150/100 mm Hg on stable antihypertensive regimen are eligible
  * History of myocardial infarction or unstable angina within the past 24 weeks
  * New York heart association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, unstable angina pectoris
  * Peripheral vascular disease ≥ grade II
* Ongoing ventricular cardiac dysrhythmias ≥ grade 2 as assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4
* History of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation > 3 beats in a row)
* Ongoing atrial fibrillation
* Pre-existing thyroid abnormality with thyroid-stimulating hormone that cannot be maintained at less than or within the normal range with medication
* Serious concurrent illness or active infection that would jeopardize the ability of the patient to receive study treatment
* Known HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-09-17 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S. Balzer-Haas, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (99):
- United States (99):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Stanford Cancer Center, Stanford, California
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - McPherson, McPherson, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Derived] Carthon BC, Kim SE, McDermott DF, Dutcher JP, Puligandla M, Manola J, Pins M, Carducci MA, Plimack ER, Appleman LJ, MacVicar GR, Kohli M, Kuzel TM, DiPaola RS, Haas NB. Results From a Randomized Phase II Trial of Sunitinib and Gemcitabine or Sunitinib in Advanced Renal Cell Carcinoma with Sarcomatoid Features: ECOG-ACRIN E1808. Clin Genitourin Cancer. 2023 Oct;21(5):546-554. doi: 10.1016/j.clgc.2023.06.012. Epub 2023 Jul 3. PMID 37455214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 patients were enrolled between June 17, 2010 and November 12, 2015. The first patient was accrued on September 17, 2010.
Period: Overall Study
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib)
Started | 47 | 40
Receipt of Protocol Therapy | 46 | 37
Treated and Eligible Patients | 45 | 37
Completed | 3 | 2
Not Completed | 44 | 38
Not completed — Progression | 24 | 25
Not completed — Adverse Event | 13 | 7
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Symptomatic deterioration | 1 | 0
Not completed — Never started treatment | 1 | 3
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib) | Total
Number analyzed (Participants) | 45 | 37 | 82
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 79] | 61 [44 to 80] | 61 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 30 | 24 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 40 | 36 | 76
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 42 | 32 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Response
Description: Response is defined as either complete response (CR, disappearance of all lesions) or partial response (PR, at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters, or persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits).
Time Frame: Assessed every 3 months for 2 years and every 6 months for year 3.
Population: Eligible and treated patients
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib)
Number analyzed (Participants) | 45 | 37
proportion of participants | 0.18 [0.11 to 0.29] | 0.11 [0.051 to 0.22]

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from randomization to progression or death, whichever occurs first. Progression is defined as follows:
  * At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  * Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Assessed every 3 months for 2 years and every 6 months for year 3.
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib)
Number analyzed (Participants) | 45 | 37
months | 4.5 [3.0 to 5.8] | 3.6 [3.0 to 7.7]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or date last known alive.
Time Frame: Assessed every 3 months for 2 years and every 6 months for year 3.
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib)
Number analyzed (Participants) | 45 | 37
months | 9.4 [7.4 to 13.0] | 7.8 [7.0 to 13.7]

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment and for 30 days after the end of treatment up to 3 years
Description: Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
Arm/Group | Arm A (Sunitinib + Gemcitabine) | Arm B (Sunitinib)
All-Cause Mortality (participants affected / at risk) | 41/47 | 31/40
Serious Adverse Events (participants affected / at risk) | 36/46 | 17/37
Other Adverse Events (participants affected / at risk) | 40/46 | 27/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sunitinib + Gemcitabine) (N=46) | Arm B (Sunitinib) (N=37)
Anemia (Blood and lymphatic system disorders) | 14 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Fatigue (General disorders) | 10 | 4
Fever (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 1 | 0
GGT increased (Investigations) | 1 | 0
Hemoglobin increased (Investigations) | 3 | 0
Lymphocyte count decreased (Investigations) | 7 | 1
Neutrophil count decreased (Investigations) | 19 | 1
Platelet count decreased (Investigations) | 6 | 1
Weight gain (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 7 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
Syncope (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 5 | 8
Hypotension (Vascular disorders) | 0 | 1
Peripheral ischemia (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Sunitinib + Gemcitabine) (N=46) | Arm B (Sunitinib) (N=37)
Anemia (Blood and lymphatic system disorders) | 19 | 3
Edema limbs (General disorders) | 3 | 1
Fatigue (General disorders) | 23 | 4
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 2 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 2 | 2
Hypothyroidism (Endocrine disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 6
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Mucositis oral (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 18 | 5
Stomach pain (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Alanine aminotransferase increased (Investigations) | 5 | 1
Alkaline phosphatase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 1
Creatinine increased (Investigations) | 4 | 3
Hemoglobin increased (Investigations) | 1 | 2
Lymphocyte count decreased (Investigations) | 4 | 4
Neutrophil count decreased (Investigations) | 14 | 3
Platelet count decreased (Investigations) | 7 | 2
White blood cell decreased (Investigations) | 11 | 5
Anorexia (Metabolism and nutrition disorders) | 7 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 7 | 5
Headache (Nervous system disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Hypertension (Vascular disorders) | 14 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT01164228/Prot_SAP_000.pdf